CLINICAL TRIAL: NCT01756859
Title: Quantitative Magnetic Resonance Imaging (MRI) Techniques in the Evaluation and Estimation of Portal Hypertension
Brief Title: MRI in Portal Hypertension
Acronym: MRQuee
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 12092
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Portal Hypertension
Keywords: Portal hypertension; HVPG; MRI
MeSH Terms: conditions — Hypertension, Portal | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood, urine and stool samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with HVPG measurements: Patients having HVPG measurements for clinical reasons will be recruited to undergo research MRI scan.
  Interventions: Procedure: MRI Scan

INTERVENTIONS:
Procedure: MRI Scan

SUMMARY:
Death from chronic liver disease has doubled in the UK over the last decade. This is largely due to the rise in liver disease from excess alcohol consumption, obesity related fatty liver disease and hepatitis B & C infections. The current 'liver tests' only identify liver injury when the damage is at an advanced stage. They neither estimate the degree of injury accurately nor help judge prognosis. The complications from chronic liver disease result mainly from raised pressures within the liver. We currently measure this pressure by passing a long catheter through the jugular vein in the neck into the liver. This invasive test does carry a small yet significant risk of complications and is not available outside specialised liver centres. Raised pressure within the liver is also associated with changes in the microorganisms within the gut. This leads to increased infective complications among patients with liver cirrhosis.

We aim to noninvasively measure the pressures within the liver using Magnetic Resonance Imaging (MRI). We will recruit 49 patients with chronic liver disease who have had liver pressure measurements as part of their routine clinical assessment. The participants will attend the Biomedical Research Unit and the MR Centre for a single 2hour visit. We will also collect blood, urine and stool samples from them.

The diagnostic accuracy of the quantitative MRI techniques will be validated against the pressures obtained via the invasive test. The quantitative MRI techniques will also correlated with biomarkers of liver injury obtained from blood and urine samples. The stool sample obtained will be used to characterise the gut microorganisms in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of more than 18 years of age.
2. Patients who have had HVPG measurements within the last 6 weeks.
3. Underlying portal hypertension due to chronic liver disease - alcoholic liver disease, non-alcoholic fatty liver disease (NAFLD), chronic hepatitis B or C and heamochromatosis.
4. Patients investigated with a clinical suspicion of portal hypertension, but have normal portal pressures on HVPG measurements.
5. Ability to consent to participate in the study.

Exclusion Criteria:

1. Patients with underlying diseases which are NOT related to alcohol excess, NAFLD, chronic hepatitis B, C or haemochromatosis.
2. Abdominal/waist circumference greater than 112 cm (44 inches) due to scanner bore constraints
3. Pregnant women.
4. Absolute contraindications for MRI. Any patient that indicates on the MR safety questionnaire that they have or suspect they may have metal in their eye(s) will require an x-ray prior to their MRI scan confirming that their eye(s) are free from metal. This will be verified using previous x-ray records. Any patient whose previous records indicate that they may have had metal in their eye(s) or any patients without any x-ray records will be x-rayed for the purposes of this study. Any patient having current metal in their eye(s), will not be given an MRI scan and therefore will not be recruited into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from liver services from Nottingham University Hospitals NHS Trust and Derby Hospitals NHS Foundation Trust. All the patients will have had HVPG measurements performed for clinical indications.
Sampling Method: Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of quantitative MR techniques in the detection and grading the degree of portal hypertension compared to HVPG measurements. | 18 months

SECONDARY OUTCOMES:
Correlation between quantitative MR techniques and serum biomarkers of fibrosis. | 18 months
Characterisation of the gut microbiota in patients with portal hypertension. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Guruprasad Aithal, Principal Investigator — NIHR Biomedical Research Unit in Gastrointestinal and Liver Diseases, Nottingham
Locations (2):
- United Kingdom (2):
  - Royal Derby Hospitals, Derby, Derby
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottingham